CLINICAL TRIAL: NCT04725539
Title: Effects of Hypoxia Pre-conditioning on Physiological Responses During Mountain Sport Activities in Persons With a History of Coronary Artery Disease
Brief Title: Hypoxia Pre-conditioning and Mountain Sport
Acronym: Hyx-PRE-Spo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Collaborators: Istituto Auxologico Italiano (Other); University of Innsbruck (Unknown); University of Giessen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HYP-P-SP
Record Dates: First submitted 2021-01-08; First posted 2021-01-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent hypoxia (IH) pre-conditioning (Experimental): The IH pre-conditioning program will be performed in a sitting position by inhaling a gas mixture with reduced O2 content via face masks.The program will include five sessions per week for 3 weeks. Each session consists of three to five hypoxic (14-10% inspired fraction of oxygen) periods, each lasting 3-5 min with 3-min normoxic intervals.
  The control setting includes breathing room air via face mask.
  Interventions: Procedure: hypoxic exposure
- Hypoxia pre-adaptation (Experimental): The hypoxia pre-adaptation program consists of sleeping 1 night at 1900m. The control setting includes sleeping 1 night close to sea level.
  Interventions: Procedure: hypoxic exposure

INTERVENTIONS:
Procedure: hypoxic exposure — Administration of different hypoxic doses.
  Intermittent hypoxia:
  days 1-5 duration of breathing periods 5*3min (FiO2 14-21%) days 8-12 duration of breathing periods 4*4min (FiO2 = 12%) and 3*3 min (FiO2 = 21%) days 15-19 duration of breathing periods 5*5min (FiO2 = 10%) and 4*3 min (FiO2 = 21%)
  one night at 1900m

SUMMARY:
Mountain sport activities as for example hiking or skiing may involve the risk of adverse health events especially in older people not accustomed to the specific mountain sport at altitude or people with pre-existing health issues. Increased activation of the sympathetic nervous system and abrupt changes in heart rate and blood pressure are thought to trigger these adverse effects. Preventive measures include regular physical activity (i.e. training) and adequate medical treatment. Hypoxia pre-adaptation (e.g., pre-adapt one night at moderate altitude) and pre-conditioning (e.g., intermittent hypoxia (IH) training), which was shown to lead to some favorable sympathetic nervous system, ventilatory and metabolic adaptations and additionally exerts anti-inflammatory action, could be hypothesized of being a further preventive measure. The aim of this research project is to investigate whether intermittent hypoxia pre-conditioning or sleeping one night at altitude (i.e., current recommendation before practicing mountain leisure sports in the elderly) is able to increase oxygen saturation during passive hypoxia exposure and during simulated hiking and skiing at altitude. Additionally, it is aimed to investigate whether such procedure reduces the physiological responses (i.e., heart rate, its variability and blood pressure (including baroreflex sensitivity) responses as well as metabolic, ventilatory, inflammatory and redox responses) during these activities.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include normally physically active males and females (age 50-70 years; New York Heart Association (NYHA) class I and II) with or without prior myocardial infarction, living <600 m.

Exclusion Criteria:

* Persons with CAD will be excluded if they will not be able to perform light to moderate exercise, or had recent myocardial infarction and/or revascularisation (< 8 weeks prior to inclusion in the study), episode of unstable angina, de-compensated heart failure, life-threatening arrhythmia, ejection fraction < 50%, known symptomatic aortic outflow obstruction, severe hypertension (>180/100 mm Hg), pulmonary hypertension or any other severe systemic non-cardiac disease. Exclusion criteria will additionally include regular smoking of more than five cigarettes per day, regular drug intake, habitual residence > 600 m and one or more overnight stay at > 1000 m during the previous 4 weeks.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Resting oxygen saturation (%) at altitude | Through study completion, an average of 1.5 years
  Resting oxygen saturation changes after the pre-conditioning and pre-adaptation program at 3000 m altitude
Oxygen saturation during exercise at altitude | Through study completion, an average of 1.5 years
  Oxygen saturation during exercise changes after the pre-conditioning and pre-adaptation program at 3000 m altitude

SECONDARY OUTCOMES:
Heart rate (bpm) responses during rest and during exercise at altitude | Through study completion, an average of 1.5 years
  Heart rate response changes after the pre-conditioning and pre-adaptation program at rest and during exercise at 3000 m altitude.
Blood pressure (mmHg) responses during rest and during exercise at altitude | Through study completion, an average of 1.5 years
  Blood pressure responses during rest and during exercise at altitude
Changes of inflammatory markers (i.e., hsCRP) from before to after the pre-conditioning and pre-adaptation program | Through study completion, an average of 1.5 years
  Inflammatory markers may change due to the programs
Changes of physiological stress markers (i.e., catecholamine) from before to after the pre-conditioning and pre-adaptation program | Through study completion, an average of 1.5 years
  Markers of physiological stress may change due to the programs
Changes in heart rate variability (HRV) from before to after the pre-conditioning and pre-adaptation program | Through study completion, an average of 1.5 years
  HRV may change due to the programs
Changes in baroreflex sensitivity (BRS) from before to after the pre-conditioning and pre-adaptation program | Through study completion, an average of 1.5 years
  BRS may change due to the programs
Changes of markers of myocardial injury (e.g., highly sensitive cardiac troponin T) from before to after the pre-conditioning and pre-adaptation program | Through study completion, an average of 1.5 years
  Markers of myocardial injury may change due to the programs

CONTACTS AND LOCATIONS:
Overall Officials: Hannes Gatterer, PhD, Principal Investigator — Institute of Mountain Emergency Medicine, EURAC Research
Locations (1):
- Eurac Research, Bolzano, BZ, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data underlying scientific publications will be stored in open repositories (accessible).
Supporting Information: Study Protocol
Time Frame: After publications
Access Criteria: The data that support the findings of this study are available from the corresponding author upon reasonable request.